CLINICAL TRIAL: NCT01170442
Title: Does Vitamin D Improve Glycemic Control in Type II DM? A Double Blind Randomized Controlled Trial
Brief Title: Does Vitamin D Improve Glycemic Control in Type II DM?
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: In adequate enrollment
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Principal Investigator, Muhammad Maher Hammami, Chairman, Department of Clinical Studies & Empirical Ethics, King Faisal Specialist Hospital & Research Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RAC 2101039
Record Dates: First submitted 2010-07-25; First posted 2010-07-27 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Diabetes Mellitus; Vitamin D Deficiency
MeSH Terms: conditions — Diabetes Mellitus; Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- vitamin D3 2000 IU (Experimental)
  Interventions: Drug: vitamin D3 2000 IU
- vitamin D3 5000 IU (Experimental)
  Interventions: Drug: vitamin D3 5000 IU
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: vitamin D3 2000 IU — vitamin D3 2000 IU orally, daily for 6 months
  Other Names: cholecalciferol
  Arms: vitamin D3 2000 IU
Drug: vitamin D3 5000 IU — vitamin D3 5000 IU orally, daily for 6 months
  Other Names: cholecalciferol
  Arms: vitamin D3 5000 IU
Drug: Placebo — placebo orally, daily for six months
  Arms: Placebo

SUMMARY:
Vitamin D status has been negatively associated with the presence of type II DM and glycemic control. However, a cause-effect relationship between vitamin D deficiency and glycemic control has not been established. The investigators plan to conduct a double blind, randomized, placebo controlled trial on the effect of vitamin D supplementation on glycemic control in Type II DM.

ELIGIBILITY:
Inclusion Criteria:

* Type II diabetics living in Riyadh area who consume no more than one serving of milk/day
* Do not take vitamin supplement
* Habitually have less than 10 hour of sun exposure per week
* Don't suffer from granulomatous conditions, liver disease, or kidney disease
* Don't take anticonvulsants, barbiturates, or steroids.
* Stable glycemic control (not more than 0.5% difference between current HA1c and a HA1c obtained 2-4 months earlier)
* Current HA1c between 6.5 and 8%, and current total 25 OH vitamin D level between 10-30 nmol/L.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2011-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Area under the curve of HA1C. | 6 months

SECONDARY OUTCOMES:
Area under the curve for BP | 6 months
area under the curve of weight | 6 months
area under the curve for 25 OH vitamin D level | 6 months
area under the curve of fasting blood glucose | 6 months
area under the curve of 2 hour post breakfast glucose | 6 months
fasting insulin to glucose ratio | 6 months
incidence of hypercalcemia | 6 months
incidence of hypercalciuria | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad M Hammami, MD, PhD, Principal Investigator — King Faisal Specialist Hospital & Research Center
Locations (1):
- King Faisal Specialist Hospital & Research Center, Riyadh, Saudi Arabia